CLINICAL TRIAL: NCT04280705
Title: A Multicenter, Adaptive, Randomized Blinded Controlled Trial of the Safety and Efficacy of Investigational Therapeutics for the Treatment of COVID-19 in Hospitalized Adults
Brief Title: Adaptive COVID-19 Treatment Trial (ACTT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-0006
Record Dates: First submitted 2020-02-20; First posted 2020-02-21 (Actual); Results first posted 2020-09-25 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2020-04

CONDITIONS: COVID-19
Keywords: Adaptive; COVID-19; Efficacy; Multicenter; novel coronavirus; Safety; ACTT
MeSH Terms: conditions — COVID-19 | interventions — remdesivir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): 200 mg of Remdesivir placebo administered intravenously on Day 1, followed by a 100 mg once-daily maintenance dose of Remdesivir placebo while hospitalized for up to a 10 days total course. n=286.
  Interventions: Other: Placebo
- Remdesivir (Experimental): 200 mg of Remdesivir administered intravenously on Day 1, followed by a 100 mg once-daily maintenance dose of Remdesivir while hospitalized for up to a 10 days total course. n=286.
  Interventions: Drug: Remdesivir

INTERVENTIONS:
Other: Placebo — The supplied placebo lyophilized formulation is identical in physical appearance to the active lyophilized formulation and contains the same inactive ingredients. Alternatively, a placebo of normal saline of equal volume may be given if there are limitations on matching placebo supplies.
  Arms: Placebo
Drug: Remdesivir — Drug Remdesivir is a single diastereomer monophosphoramidate prodrug designed for the intracellular delivery of a modified adenine nucleoside analog GS-441524. In addition to the active ingredient, the lyophilized formulation of Remdesivir contains the following inactive ingredients: water for injection, sulfobutylether beta-cyclodextrin sodium (SBECD), and hydrochloric acid and/or sodium hydroxide.
  Arms: Remdesivir

SUMMARY:
This study is an adaptive, randomized, double-blind, placebo-controlled trial to evaluate the safety and efficacy of novel therapeutic agents in hospitalized adults diagnosed with COVID-19. The study is a multicenter trial that will be conducted in up to approximately 100 sites globally. The study will compare different investigational therapeutic agents to a control arm. There will be interim monitoring to introduce new arms and allow early stopping for futility, efficacy, or safety. If one therapy proves to be efficacious, then this treatment may become the control arm for comparison(s) with new experimental treatment(s). Any such change would be accompanied by an updated sample size. Because background standards of supportive care may evolve/improve over time as more is learned about successful management of COVID-19, comparisons of safety and efficacy will be based on data from concurrently randomized subjects. An independent Data and Safety Monitoring Board (DSMB) will actively monitor interim data to make recommendations about early study closure or changes to study arms. To evaluate the clinical efficacy, as assessed by time to recovery, of different investigational therapeutics as compared to the control arm.

DETAILED DESCRIPTION:
This study is an adaptive, randomized, double-blind, placebo-controlled trial to evaluate the safety and efficacy of novel therapeutic agents in hospitalized adults diagnosed with COVID-19. The study is a multicenter trial that will be conducted in up to approximately 100 sites globally. The study will compare different investigational therapeutic agents to a control arm. There will be interim monitoring to introduce new arms and allow early stopping for futility, efficacy, or safety. If one therapy proves to be efficacious, then this treatment may become the control arm for comparison(s) with new experimental treatment(s). Any such change would be accompanied by an updated sample size. Because background standards of supportive care may evolve/improve over time as more is learned about successful management of COVID-19, comparisons of safety and efficacy will be based on data from concurrently randomized subjects. An independent Data and Safety Monitoring Board (DSMB) will actively monitor interim data to make recommendations about early study closure or changes to study arms.

The initial sample size is projected to be 572 subjects to achieve 400 subjects with a "recovered" status (per the primary objective). The primary analysis will be based on those subjects enrolled in order to 400 recoveries. An additional analysis of the moderate severity subgroup (those with baseline status of "Hospitalized, requiring supplemental oxygen" or "Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care") is also of public health importance. Hence, enrollment will be permitted until the date of April 20, 2020 to ensure 400 recoveries and provide additional data about this important subgroup. With recent enrollment rates, the total sample size may be 600 to over 800.

Subjects will be assessed daily while hospitalized. If the subjects are discharged from the hospital, they will have a study visit at Days 15, 22, and 29 as an outpatient. For discharged subjects, it is preferred that the Day 15 and 29 visits are in person to obtain safety laboratory tests and OP swab and blood (serum only) samples for secondary research as well as clinical outcome data. However, infection control or other restrictions may limit the ability of the subject to return to the clinic. In this case, Day 15 and 29 visits may be conducted by phone, and only clinical data will be obtained. The Day 22 visit does not have laboratory tests or collection of samples and may also be conducted by phone.

All subjects will undergo a series of efficacy, safety, and laboratory assessments. Safety laboratory tests and blood (serum and plasma) research samples and oropharyngeal (OP) swabs will be obtained on Days 1 (prior to infusion) and Days 3, 5, 8, and 11 (while hospitalized). OP swabs and blood (serum only) plus safety laboratory tests will be collected on Day 15 and 29 (if the subject attends an in-person visit or are still hospitalized).

The primary outcome is time to recovery by Day 29. A key secondary outcome evaluates treatment-related improvements in the 8-point ordinal scale at Day 15. As little is known about the clinical course of COVID-19, a pilot study will be used for a blinded sample size reassessment.

Contacts:

20-0006 Central Contact

Telephone: 1 (301) 7617948

Email: DMIDClinicalTrials@niaid.nih.gov

ELIGIBILITY:
Inclusion Criteria:

1. Admitted to a hospital with symptoms suggestive of COVID-19 infection.
2. Subject (or legally authorized representative) provides informed consent prior to initiation of any study procedures.
3. Subject (or legally authorized representative) understands and agrees to comply with planned study procedures.
4. Male or non-pregnant female adult > / = 18 years of age at time of enrollment.
5. Has laboratory-confirmed SARS-CoV-2 infection as determined by polymerase chain reaction (PCR) or other commercial or public health assay in any specimen, as documented by either or the following:

   1. PCR positive in sample collected < 72 hours prior to randomization; OR

      Exclusion Criteria:
   2. PCR positive in sample collected >/= 72 hours prior to randomization, documented inability to obtain a repeat sample (e.g. due to lack of testing supplies, limited testing capacity, results taking >24 hours, etc.) AND progressive disease suggestive of ongoing SARS-CoV-2 infection.
6. Illness of any duration, and at least one of the following:

   1. Radiographic infiltrates by imaging (chest x-ray, CT scan, etc.), OR
   2. SpO2 < / = 94% on room air, OR
   3. Requiring supplemental oxygen, OR
   4. Requiring mechanical ventilation.
7. Women of childbearing potential must agree to either abstinence or use at least one primary form of contraception not including hormonal contraception from the time of screening through Day 29.
8. Agrees to not participate in another clinical trial for the treatment of COVID-19 or SARS-CoV-2 through Day 29.

Exclusion Criteria:

1. Alanine Transaminase (ALT) or Aspartate Transaminase (AST) > 5 times the upper limit of normal.
2. Estimated glomerular filtration rate (eGFR) < 30 ml/min (including patients receiving hemodialysis or hemofiltration).
3. Pregnancy or breast feeding.
4. Anticipated discharge from the hospital or transfer to another hospital which is not a study site within 72 hours.
5. Allergy to any study medication.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1062 (Actual)
Dates: Start 2020-02-21 (Actual); Primary Completion 2020-05-21 (Actual); Study Completion 2020-05-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (60):
- United States (41):
  - University of Alabama at Birmingham School of Medicine - Infectious Disease, Birmingham, Alabama
  - University of California San Diego Health - Jacobs Medical Center, La Jolla, California
  - University of California Los Angeles Medical Center - Westwood Clinic, Los Angeles, California
  - University of California Irvine Medical Center - Infectious Disease, Orange, California
  - VA Palo Alto Health Care System - Infectious Diseases, Palo Alto, California
  - University of California Davis Medical Center - Internal Medicine - Infectious Disease, Sacramento, California
  - Naval Medical Center San Diego - Infectious Disease Clinic, San Diego, California
  - University of California San Francisco - Zuckerberg San Francisco General Hospital - Division of Human Immunodeficiency Virus, Infectious Disease, and Global Medicine, San Francisco, California
  - Stanford University - Stanford Hospital and Clinics - Pediatrics - Infectious Diseases, Stanford, California
  - Cedars Sinai Medical Center, West Hollywood, California
  - Denver Health Division of Hospital Medicine - Main Campus, Denver, Colorado
  - Emory Vaccine Center - The Hope Clinic, Decatur, Georgia
  - Northwestern Hospital - Infectious Disease, Chicago, Illinois
  - University of Illinois at Chicago College of Medicine - Division of Infectious Diseases, Chicago, Illinois
  - Southeast Louisiana Veterans Health Care System - Section of Infectious Diseases, New Orleans, Louisiana
  - University of Maryland School of Medicine - Center for Vaccine Development - Baltimore, Baltimore, Maryland
  - Johns Hopkins Hospital - Medicine - Infectious Diseases, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - National Institutes of Health - Clinical Center, National Institute of Allergy and Infectious Diseases Laboratory Of Immunoregulation, Clinical Research Section, Bethesda, Maryland
  - Massachusetts General Hospital - Infectious Diseases, Boston, Massachusetts
  - University of Massachusetts Medical School - Infectious Diseases and Immunology, Worcester, Massachusetts
  - University of Minnesota Medical Center, Fairview - Infectious Diseases and International Medicine, Minneapolis, Minnesota
  - Saint Louis University - Center for Vaccine Development, St Louis, Missouri
  - University of Nebraska Medical Center - Infectious Diseases, Omaha, Nebraska
  - New York University School of Medicine - Langone Medical Center - Microbiology - Parasitology, New York, New York
  - University of Rochester Medical Center - Vaccine Research Unit, Rochester, New York
  - Montefiore Medical Center - Infectious Diseases, The Bronx, New York
  - Duke Human Vaccine Institute - Duke Vaccine and Trials Unit, Durham, North Carolina
  - Penn State Health Milton S. Hershey Medical Center - Division of Infectious Diseases, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania - Infectious Diseases, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center - Infectious Diseases, Nashville, Tennessee
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch - Division of Infectious Disease, Galveston, Texas
  - Baylor College of Medicine - Molecular Virology and Microbiology, Houston, Texas
  - University of Texas Health Science Center at San Antonio - Infectious Diseases, San Antonio, Texas
  - University of Virginia - Acute Care Surgery, Charlottesville, Virginia
  - Naval Medical Center Portsmouth - Infectious Disease Division, Portsmouth, Virginia
  - EvergreenHealth Infectious Disease Service, Kirkland, Washington
  - The University of Washington - Virology Research Clinic, Seattle, Washington
  - Providence Sacred Heart Medical Center, Spokane, Washington
  - Madigan Army Medical Center - Infectious Disease Clinic, Tacoma, Washington
- University of Copenhagen - Centre of Excellence for Health, Immunity and Infections (CHIP) - Department of Infectious Diseases, Copenhagen, Denmark
- Germany (3):
  - Universitatsklinikum Bonn, Medizinische Klinik I - Bereich Infektiologie/HIV der Medizinischen Klinik, Bonn, North Rhine-Westphalia
  - Universitatsklinikum Koeln Klinik I fur Innere Medizin Klinisches Studienzentrum fur Infektiologie I, Cologne
  - Universitätsklinikum Frankfurt -Medizinische Klinik II - Infektiologie, Frankfurt
- Greece (2):
  - AHEPA University Hospital - 1st Department of Internal Medicine, Thessaloniki, Central Macedonia
  - Medical School of Athens University - Evangelismos Hospital - Department of Critical Care and Pulmonary Services, Athens
- National Center for Global Health and Medicine Hospital - Disease Control and Prevention Center, Tokyo, Japan
- Mexico (2):
  - Instituto Nacional de Ciencias Medicas y Nutrición Salvador Zubirán - Departamento de Infectologia, Mexico City
  - Instituto Nacional de Enfermedades Respiratorias (INER) - Ismael Cosío Villegas, Mexico City
- National Centre for Infectious Diseases, Singapore, Singapore
- South Korea (2):
  - Seoul National University Bundang Hospital - Division of Infectious Diseases, Bundang-gu Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul, Jongno-gu
- Spain (2):
  - Hospital Clinic Barcelona, Servicio de Salud Internacional, Barcelona, Catalonia
  - Hospital Germans Trias i Pujol - Servei Malalties Infeccioses, Barcelona, Catalonia
- United Kingdom (5):
  - Royal Sussex County Hospital - Department of Intensive Care Medicine, East Sussex, Brighton
  - Saint Thomas' Hospital - Directorate of Infection, London, London, City of
  - Royal Victoria Infirmary - Department of Infectious Diseases, Level 6, Ward 19, Newcastle Upon Tyne
  - St. James's University Hospital - Infectious Diseases, Leeds, West Yorkshire
  - John Radcliffe Hospital, Headington, Oxford

REFERENCES:
- [Derived] Singh K, Rubenstein K, Callier V, Shaw-Saliba K, Rupert A, Dewar R, Laverdure S, Highbarger H, Lallemand P, Huang ML, Jerome KR, Sampoleo R, Mills MG, Greninger AL, Juneja K, Porter D, Benson CA, Dempsey W, El Sahly HM, Focht C, Jilg N, Paules CI, Rapaka RR, Uyeki TM, Clifford Lane H, Beigel J, Dodd LE; Adaptive COVID-19 Treatment Trial (ACTT-1) Study Group Members. SARS-CoV-2 RNA and Nucleocapsid Antigen Are Blood Biomarkers Associated With Severe Disease Outcomes That Improve in Response to Remdesivir. J Infect Dis. 2024 Sep 23;230(3):624-634. doi: 10.1093/infdis/jiae198. PMID 38657001
- [Derived] Hedskog C, Rodriguez L, Roychoudhury P, Huang ML, Jerome KR, Hao L, Ireton RC, Li J, Perry JK, Han D, Camus G, Greninger AL, Gale M Jr, Porter DP. Viral Resistance Analyses From the Remdesivir Phase 3 Adaptive COVID-19 Treatment Trial-1 (ACTT-1). J Infect Dis. 2023 Nov 2;228(9):1263-1273. doi: 10.1093/infdis/jiad270. PMID 37466213
- [Derived] Grundeis F, Ansems K, Dahms K, Thieme V, Metzendorf MI, Skoetz N, Benstoem C, Mikolajewska A, Griesel M, Fichtner F, Stegemann M. Remdesivir for the treatment of COVID-19. Cochrane Database Syst Rev. 2023 Jan 25;1(1):CD014962. doi: 10.1002/14651858.CD014962.pub2. PMID 36695483
- [Derived] Potter GE, Bonnett T, Rubenstein K, Lindholm DA, Rapaka RR, Doernberg SB, Lye DC, Mularski RA, Hynes NA, Kline S, Paules CI, Wolfe CR, Frank MG, Rouphael NG, Deye GA, Sweeney DA, Colombo RE, Davey RT Jr, Mehta AK, Whitaker JA, Castro JG, Amin AN, Colombo CJ, Levine CB, Jain MK, Maves RC, Marconi VC, Grossberg R, Hozayen S, Burgess TH, Atmar RL, Ganesan A, Gomez CA, Benson CA, Lopez de Castilla D, Ahuja N, George SL, Nayak SU, Cohen SH, Lalani T, Short WR, Erdmann N, Tomashek KM, Tebas P. Temporal Improvements in COVID-19 Outcomes for Hospitalized Adults: A Post Hoc Observational Study of Remdesivir Group Participants in the Adaptive COVID-19 Treatment Trial. Ann Intern Med. 2022 Dec;175(12):1716-1727. doi: 10.7326/M22-2116. Epub 2022 Nov 29. PMID 36442063
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343
- [Derived] Ansems K, Grundeis F, Dahms K, Mikolajewska A, Thieme V, Piechotta V, Metzendorf MI, Stegemann M, Benstoem C, Fichtner F. Remdesivir for the treatment of COVID-19. Cochrane Database Syst Rev. 2021 Aug 5;8(8):CD014962. doi: 10.1002/14651858.CD014962. PMID 34350582
- [Derived] Sultana J, Crisafulli S, Gabbay F, Lynn E, Shakir S, Trifiro G. Challenges for Drug Repurposing in the COVID-19 Pandemic Era. Front Pharmacol. 2020 Nov 6;11:588654. doi: 10.3389/fphar.2020.588654. eCollection 2020. PMID 33240091
- [Derived] Maleszewski JJ, Young PM, Ackerman MJ, Halushka MK. Urgent Need for Studies of the Late Effects of SARS-CoV-2 on the Cardiovascular System. Circulation. 2021 Mar 30;143(13):1271-1273. doi: 10.1161/CIRCULATIONAHA.120.051362. Epub 2020 Sep 24. No abstract available. PMID 32969710
- [Derived] Beigel JH, Tomashek KM, Dodd LE, Mehta AK, Zingman BS, Kalil AC, Hohmann E, Chu HY, Luetkemeyer A, Kline S, Lopez de Castilla D, Finberg RW, Dierberg K, Tapson V, Hsieh L, Patterson TF, Paredes R, Sweeney DA, Short WR, Touloumi G, Lye DC, Ohmagari N, Oh MD, Ruiz-Palacios GM, Benfield T, Fatkenheuer G, Kortepeter MG, Atmar RL, Creech CB, Lundgren J, Babiker AG, Pett S, Neaton JD, Burgess TH, Bonnett T, Green M, Makowski M, Osinusi A, Nayak S, Lane HC; ACTT-1 Study Group Members. Remdesivir for the Treatment of Covid-19 - Final Report. N Engl J Med. 2020 Nov 5;383(19):1813-1826. doi: 10.1056/NEJMoa2007764. Epub 2020 Oct 8. PMID 32445440

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the participating sites from those admitted with symptoms of COVID-19 confirmed by PCR. Enrollment occurred between 21FEB2020 and 20APR2020.
Groups:
- Placebo: 200 mg of Remdesivir placebo administered intravenously on Day 1, followed by a 100 mg once-daily maintenance dose of Remdesivir placebo while hospitalized for up to a 10 days total course.
  Placebo: The supplied placebo lyophilized formulation is identical in physical appearance to the active lyophilized formulation and contains the same inactive ingredients. Alternatively, a placebo of normal saline of equal volume may be given if there are limitations on matching placebo supplies.
- Remdesivir: 200 mg of Remdesivir administered intravenously on Day 1, followed by a 100 mg once-daily maintenance dose of Remdesivir while hospitalized for up to a 10 days total course.
  Remdesivir: Drug Remdesivir is a single diastereomer monophosphoramidate prodrug designed for the intracellular delivery of a modified adenine nucleoside analog GS-441524. In addition to the active ingredient, the lyophilized formulation of Remdesivir contains the following inactive ingredients: water for injection, sulfobutylether beta-cyclodextrin sodium (SBECD), and hydrochloric acid and/or sodium hydroxide.
Period: Overall Study
Arm/Group | Placebo | Remdesivir
Started | 521 | 541
Received Treatment | 517 | 531
Completed | 508 | 517
Not Completed | 13 | 24
Not completed — Enrolled but not treated | 4 | 10
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 7 | 9
Not completed — Adverse Event | 0 | 4
Not completed — Transferred to another hospital | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: 200 mg of Remdesivir placebo administered intravenously on Day 1, followed by a 100 mg once-daily maintenance dose of Remdesivir placebo while hospitalized for up to a 10 days total course.
- Remdesivir: 200 mg of Remdesivir administered intravenously on Day 1, followed by a 100 mg once-daily maintenance dose of Remdesivir while hospitalized for up to a 10 days total course.
- Total: Total of all reporting groups
Arm/Group | Placebo | Remdesivir | Total
Number analyzed (Participants) | 521 | 541 | 1062
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 324 | 354 | 678
  >=65 years | 197 | 187 | 384
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (15.4) | 58.6 (14.6) | 58.9 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 189 | 189 | 378
  Male | 332 | 352 | 684
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 116 | 134 | 250
  Not Hispanic or Latino | 373 | 382 | 755
  Unknown or Not Reported | 32 | 25 | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 4 | 7
  Asian | 56 | 79 | 135
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
  Black or African American | 117 | 109 | 226
  White | 287 | 279 | 566
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 55 | 66 | 121
Region of Enrollment [Number; unit: participants]
  Greece | 19 | 14 | 33
  South Korea | 12 | 9 | 21
  Singapore | 7 | 9 | 16
  United States | 410 | 427 | 837
  Japan | 7 | 8 | 15
  Denmark | 21 | 22 | 43
  Mexico | 6 | 4 | 10
  United Kingdom | 21 | 25 | 46
  Germany | 6 | 7 | 13
  Spain | 12 | 16 | 28
Disease severity [Count of Participants; unit: Participants] — Mild-moderate disease: SpO2 > 94% and respiratory rate < 24 breaths/min without supplemental oxygen.
  Severe disease: requiring mechanical ventilation, requiring oxygen, a SpO2 = 94% on room air, or tachypnea (respiratory rate = 24 breaths/min).
  Participants
    Mild-to-moderate disease severity | 50 | 55 | 105
    Severe disease severity | 471 | 486 | 957

OUTCOME MEASURES:

1. Primary Outcome: Time to Recovery
Description: Day of recovery is defined as the first day on which the subject satisfies one of the following three categories from the ordinal scale: 1) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 2) Not hospitalized, limitation on activities and/or requiring home oxygen; 3) Not hospitalized, no limitations on activities.
Time Frame: Day 1 through Day 29
Population: The intent-to-treat (ITT) population includes all participants who were randomized
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo | Remdesivir
Number analyzed (Participants) | 521 | 541
Days | 15 [13 to 18] | 10 [9 to 11]
Statistical Analysis 1: Comparison: Placebo vs Remdesivir; Test type: Superiority; p < 0.001, Log Rank; Cox Proportional Hazard = 1.29, 95% CI 2-sided [1.12 to 1.49]

2. Secondary Outcome: Change From Baseline in Alanine Transaminase (ALT)
Description: Blood to evaluate ALT was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: The safety population includes all treated participants with available data at baseline and the post baseline assessment point, analyzed as treated.
Measure: Mean (Standard Deviation); unit: Units/Liter (U/L)
Arm/Group | Placebo | Remdesivir
Number analyzed (Participants) | 463 | 465
Units/Liter (U/L)
  Day 3 | 14.3 (88) | 2.9 (31.5)
  Day 5: number analyzed (Participants) | 403 | 398
  Day 5 | 23.1 (70.6) | 10.8 (55.8)
  Day 8: number analyzed (Participants) | 327 | 296
  Day 8 | 24.2 (79.7) | 8.9 (54.2)
  Day 11: number analyzed (Participants) | 257 | 227
  Day 11 | 27.7 (89.8) | 3.4 (48.4)
  Day 15: number analyzed (Participants) | 242 | 257
  Day 15 | 28.1 (110.1) | 1.7 (47.4)
  Day 29: number analyzed (Participants) | 180 | 220
  Day 29 | -3.9 (62.2) | -6.8 (43.7)

3. Secondary Outcome: Change From Baseline in Aspartate Transaminase (AST)
Description: Blood to evaluate AST was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units/Liter (U/L)
Arm/Group | Placebo | Remdesivir
Number analyzed (Participants) | 438 | 445
Units/Liter (U/L)
  Day 3 | 13.7 (90.7) | -2.0 (29.1)
  Day 5: number analyzed (Participants) | 384 | 380
  Day 5 | 12.8 (66.2) | 6.0 (58.9)
  Day 8: number analyzed (Participants) | 315 | 285
  Day 8 | 13.1 (114.6) | 1.1 (55.9)
  Day 11: number analyzed (Participants) | 247 | 219
  Day 11 | 11.5 (78.8) | -0.3 (51.7)
  Day 15: number analyzed (Participants) | 236 | 248
  Day 15 | 4.2 (73.0) | -2.3 (60.4)
  Day 29: number analyzed (Participants) | 170 | 208
  Day 29 | -18.4 (47.2) | -14.0 (52.2)

4. Secondary Outcome: Change From Baseline in Creatinine
Description: Blood to evaluate serum creatinine was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milligrams/deciliter (mg/dL)
Arm/Group | Placebo | Remdesivir
Number analyzed (Participants) | 475 | 482
milligrams/deciliter (mg/dL)
  Day 3 | 0.037 (0.517) | 0.038 (0.569)
  Day 5: number analyzed (Participants) | 418 | 411
  Day 5 | -0.695 (17.552) | 0.075 (0.762)
  Day 8: number analyzed (Participants) | 335 | 309
  Day 8 | -0.882 (19.637) | 0.158 (0.951)
  Day 11: number analyzed (Participants) | 269 | 234
  Day 11 | 1.173 (15.440) | 0.236 (1.057)
  Day 15: number analyzed (Participants) | 249 | 262
  Day 15 | -1.239 (22.755) | 0.319 (2.147)
  Day 29: number analyzed (Participants) | 189 | 229
  Day 29 | -1.863 (26.093) | 0.075 (0.644)

5. Secondary Outcome: Change From Baseline in Glucose
Description: Blood to evaluate serum glucose was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Remdesivir
Number analyzed (Participants) | 456 | 459
mg/dL
  Day 3 | -0.2 (53.4) | -3.0 (49.4)
  Day 5: number analyzed (Participants) | 407 | 395
  Day 5 | 6.3 (60.2) | 2.1 (63.8)
  Day 8: number analyzed (Participants) | 323 | 301
  Day 8 | 2.2 (73.3) | 3.2 (68.0)
  Day 11: number analyzed (Participants) | 260 | 228
  Day 11 | 1.0 (70.1) | -0.1 (77.4)
  Day 15: number analyzed (Participants) | 241 | 250
  Day 15 | -2.8 (64.4) | -2.9 (75.4)
  Day 29: number analyzed (Participants) | 180 | 219
  Day 29 | -13.5 (96.8) | -11.7 (75.4)

6. Secondary Outcome: Change From Baseline in Hemoglobin
Description: Blood to evaluate hemoglobin was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: grams/deciliter (g/dL)
Arm/Group | Placebo | Remdesivir
Number analyzed (Participants) | 475 | 475
grams/deciliter (g/dL)
  Day 3 | -0.52 (1.10) | -0.69 (5.36)
  Day 5: number analyzed (Participants) | 420 | 406
  Day 5 | -0.83 (1.22) | -0.99 (5.83)
  Day 8: number analyzed (Participants) | 334 | 310
  Day 8 | -1.22 (1.42) | -0.49 (6.54)
  Day 11: number analyzed (Participants) | 269 | 230
  Day 11 | -1.66 (1.67) | -1.29 (1.93)
  Day 15: number analyzed (Participants) | 253 | 260
  Day 15 | -1.51 (2.02) | -1.02 (3.04)
  Day 29: number analyzed (Participants) | 189 | 227
  Day 29 | -1.02 (2.38) | -1.21 (7.91)

7. Secondary Outcome: Change From Baseline in Platelets
Description: Blood to evaluate platelets was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^9 cells/liter
Arm/Group | Placebo | Remdesivir
Number analyzed (Participants) | 471 | 474
10^9 cells/liter
  Day 3 | 39.3 (60.0) | 46.0 (62.6)
  Day 5: number analyzed (Participants) | 419 | 403
  Day 5 | 76.5 (100.5) | 90.1 (99.9)
  Day 8: number analyzed (Participants) | 332 | 308
  Day 8 | 111.8 (137.4) | 130.8 (128.1)
  Day 11: number analyzed (Participants) | 269 | 229
  Day 11 | 109.3 (149.3) | 101.0 (145.0)
  Day 15: number analyzed (Participants) | 252 | 258
  Day 15 | 96.5 (154.2) | 71.1 (133.3)
  Day 29: number analyzed (Participants) | 189 | 224
  Day 29 | 32.7 (124.2) | 39.6 (107.4)

8. Secondary Outcome: Change From Baseline in Prothrombin Time (PT)
Description: Blood to evaluate PT was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Placebo | Remdesivir
Number analyzed (Participants) | 339 | 352
seconds
  Day 3 | -0.18 (4.28) | 0.44 (5.22)
  Day 5: number analyzed (Participants) | 296 | 306
  Day 5 | -0.30 (4.72) | 1.15 (5.72)
  Day 8: number analyzed (Participants) | 246 | 234
  Day 8 | 0.01 (2.59) | 1.43 (3.89)
  Day 11: number analyzed (Participants) | 199 | 182
  Day 11 | 0.86 (7.85) | 1.88 (5.68)
  Day 15: number analyzed (Participants) | 176 | 193
  Day 15 | 0.34 (4.33) | -0.03 (4.25)
  Day 29: number analyzed (Participants) | 134 | 163
  Day 29 | -0.28 (3.20) | -0.63 (3.37)

9. Secondary Outcome: Change From Baseline in Total Bilirubin
Description: Blood to evaluate total bilirubin was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Remdesivir
Number analyzed (Participants) | 451 | 456
mg/dL
  Day 3 | 0.08 (1.25) | -0.04 (0.75)
  Day 5: number analyzed (Participants) | 394 | 389
  Day 5 | 0.58 (4.13) | -0.03 (1.03)
  Day 8: number analyzed (Participants) | 315 | 288
  Day 8 | 0.22 (2.56) | 0.01 (1.38)
  Day 11: number analyzed (Participants) | 247 | 220
  Day 11 | 0.23 (2.79) | 0.07 (1.48)
  Day 15: number analyzed (Participants) | 237 | 254
  Day 15 | 0.00 (1.80) | 0.09 (1.54)
  Day 29: number analyzed (Participants) | 178 | 216
  Day 29 | -0.17 (1.65) | -0.12 (1.77)

10. Secondary Outcome: Change From Baseline in White Blood Cell Count (WBC)
Description: Blood to evaluate WBC was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^9 cells/liter
Arm/Group | Placebo | Remdesivir
Number analyzed (Participants) | 474 | 475
10^9 cells/liter
  Day 3 | 18.691 (424.837) | -18.970 (301.944)
  Day 5: number analyzed (Participants) | 419 | 405
  Day 5 | 9.886 (566.175) | -28.209 (412.615)
  Day 8: number analyzed (Participants) | 333 | 310
  Day 8 | 27.223 (479.095) | -45.997 (602.461)
  Day 11: number analyzed (Participants) | 268 | 230
  Day 11 | 1.967 (16.042) | -34.702 (574.065)
  Day 15: number analyzed (Participants) | 252 | 260
  Day 15 | 56.311 (620.551) | -70.884 (600.011)
  Day 29: number analyzed (Participants) | 189 | 226
  Day 29 | -0.898 (17.801) | 0.251 (3.987)

11. Secondary Outcome: Change From Baseline in Neutrophils
Description: Blood to evaluate neutrophils was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^9 cells/liter
Arm/Group | Placebo | Remdesivir
Number analyzed (Participants) | 463 | 459
10^9 cells/liter
  Day 3 | 9.429 (260.345) | -8.093 (135.068)
  Day 5: number analyzed (Participants) | 406 | 389
  Day 5 | 4.177 (362.782) | -15.067 (216.532)
  Day 8: number analyzed (Participants) | 317 | 298
  Day 8 | 17.916 (305.321) | -28.179 (365.099)
  Day 11: number analyzed (Participants) | 257 | 220
  Day 11 | 3.010 (27.502) | -21.773 (354.025)
  Day 15: number analyzed (Participants) | 241 | 253
  Day 15 | 36.024 (389.093) | -39.988 (333.088)
  Day 29: number analyzed (Participants) | 177 | 218
  Day 29 | -1.269 (7.160) | -0.840 (3.666)

12. Secondary Outcome: Change From Baseline in Lymphocytes
Description: Blood to evaluate lymphocytes was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^9 cells/liter
Arm/Group | Placebo | Remdesivir
Number analyzed (Participants) | 463 | 459
10^9 cells/liter
  Day 3 | 5.883 (118.740) | -7.847 (131.548)
  Day 5: number analyzed (Participants) | 406 | 389
  Day 5 | 4.064 (141.580) | -11.723 (167.428)
  Day 8: number analyzed (Participants) | 317 | 299
  Day 8 | 8.006 (137.149) | -15.455 (194.111)
  Day 11: number analyzed (Participants) | 257 | 220
  Day 11 | 0.393 (1.371) | -12.016 (183.060)
  Day 15: number analyzed (Participants) | 241 | 253
  Day 15 | 14.793 (159.583) | -23.836 (218.653)
  Day 29: number analyzed (Participants) | 177 | 218
  Day 29 | 0.668 (1.406) | 0.743 (0.664)

13. Secondary Outcome: Change From Baseline in Monocytes
Description: Blood to evaluate monocytes was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^9 cells/liter
Arm/Group | Placebo | Remdesivir
Number analyzed (Participants) | 463 | 458
10^9 cells/liter
  Day 3 | 2.448 (41.304) | -2.940 (46.752)
  Day 5: number analyzed (Participants) | 406 | 388
  Day 5 | 1.498 (57.686) | -2.628 (39.329)
  Day 8: number analyzed (Participants) | 316 | 299
  Day 8 | 2.324 (36.626) | -3.645 (48.636)
  Day 11: number analyzed (Participants) | 257 | 220
  Day 11 | 0.383 (0.744) | -2.539 (43.454)
  Day 15: number analyzed (Participants) | 241 | 253
  Day 15 | 6.475 (69.019) | -8.738 (74.365)
  Day 29: number analyzed (Participants) | 177 | 218
  Day 29 | 0.125 (0.485) | 0.117 (0.340)

14. Secondary Outcome: Change From Baseline in Basophils
Description: Blood to evaluate basophils was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^9 cells/liter
Arm/Group | Placebo | Remdesivir
Number analyzed (Participants) | 455 | 452
10^9 cells/liter
  Day 3 | 0.020 (0.257) | 0.005 (0.043)
  Day 5: number analyzed (Participants) | 394 | 380
  Day 5 | 0.038 (0.501) | 0.005 (0.370)
  Day 8: number analyzed (Participants) | 309 | 293
  Day 8 | 0.196 (3.132) | 0.005 (0.368)
  Day 11: number analyzed (Participants) | 253 | 218
  Day 11 | 0.024 (0.042) | 0.028 (0.053)
  Day 15: number analyzed (Participants) | 235 | 248
  Day 15 | 0.158 (1.913) | -0.058 (1.028)
  Day 29: number analyzed (Participants) | 176 | 216
  Day 29 | 0.040 (0.073) | 0.029 (0.054)

15. Secondary Outcome: Change From Baseline in Eosinophils
Description: Blood to evaluate eosinophils was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^9 cells/liter
Arm/Group | Placebo | Remdesivir
Number analyzed (Participants) | 456 | 455
10^9 cells/liter
  Day 3 | 0.634 (10.614) | 0.016 (0.727)
  Day 5: number analyzed (Participants) | 397 | 387
  Day 5 | 0.666 (11.977) | -0.066 (2.807)
  Day 8: number analyzed (Participants) | 311 | 293
  Day 8 | 0.596 (8.875) | -0.221 (4.108)
  Day 11: number analyzed (Participants) | 254 | 218
  Day 11 | 0.093 (0.190) | -0.088 (2.973)
  Day 15: number analyzed (Participants) | 237 | 251
  Day 15 | 1.992 (20.365) | -0.420 (5.378)
  Day 29: number analyzed (Participants) | 176 | 217
  Day 29 | 0.241 (0.324) | 0.211 (0.267)

16. Secondary Outcome: Change in National Early Warning Score (NEWS) From Baseline
Description: The NEW score has demonstrated an ability to discriminate patients at risk of poor outcomes. This score is based on 7 clinical parameters (respiration rate, oxygen saturation, any supplemental oxygen, temperature, systolic blood pressure, heart rate, level of consciousness). The NEW Score is being used as an efficacy measure. The minimum score is 0, representing the better outcome, and the maximum value is 19, representing the worse outcome.
Time Frame: Days 1, 3, 5, 8, 11, 15, 22, and 29
Population: The intent-to-treat (ITT) population includes all participants who were randomized with data at baseline and at each timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Remdesivir
Number analyzed (Participants) | 499 | 502
units on a scale
  Day 3 | 0.1 (2.8) | -0.3 (2.6)
  Day 5: number analyzed (Participants) | 447 | 438
  Day 5 | 0.3 (3.3) | -0.4 (2.9)
  Day 8: number analyzed (Participants) | 348 | 321
  Day 8 | -0.3 (3.8) | -0.5 (3.2)
  Day 11: number analyzed (Participants) | 291 | 254
  Day 11 | -0.3 (4.1) | -0.5 (3.5)
  Day 15: number analyzed (Participants) | 290 | 301
  Day 15 | -1.4 (4.2) | -1.7 (3.6)
  Day 22: number analyzed (Participants) | 151 | 120
  Day 22 | -1.4 (4.0) | -1.7 (4.1)
  Day 29: number analyzed (Participants) | 221 | 251
  Day 29 | -3.2 (4.0) | -3.3 (3.2)

17. Secondary Outcome: Percentage of Participants at Each Clinical Status Using Ordinal Scale at Day 1
Description: The ordinal scale is an assessment of the clinical status at the first assessment of a given study day. The scale is as follows: 8) Death; 7) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 6) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 5) Hospitalized, requiring supplemental oxygen; 4) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 3) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 2) Not hospitalized, limitation on activities and/or requiring home oxygen; 1) Not hospitalized, no limitations on activities.
Time Frame: Day 1
Population: The intent-to-treat (ITT) population includes all participants who were randomized
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Remdesivir
Number analyzed (Participants) | 521 | 541
percentage of participants
  Death at or before study Visit | 0 [0 to 1] | 0 [0 to 1]
  Hospitalized, on invasive mech. vent. or ECMO | 30 [26 to 34] | 24 [21 to 28]
  Hospitalized, on non-invasive vent./high flow O2 | 19 [16 to 22] | 18 [15 to 21]
  Hospitalized, requiring supplemental oxygen | 39 [35 to 43] | 43 [39 to 47]
  Hospitalized, not on O2, requiring ongoing care | 12 [10 to 15] | 14 [11 to 17]
  Hospitalized, not requiring O2, no longer req care | 0 [0 to 1] | 0 [0 to 1]
  Not hospitalized, limit on activities/req home O2 | 0 [0 to 1] | 0 [0 to 1]
  Not hospitalized, no limitations on activities | 0 [0 to 1] | 0 [0 to 1]
  No clinical status score reported - Hospitalized | 0 [0 to 1] | 1 [0 to 2]
  No clinical status score reported - Discharged | 0 [0 to 1] | 0 [0 to 1]
  No clinical status score reported - Discontinued | 1 [0 to 2] | 1 [0 to 2]

18. Secondary Outcome: Percentage of Participants at Each Clinical Status Using Ordinal Scale at Day 3
Description: as for outcome 17
Time Frame: Day 3
Population: The intent-to-treat (ITT) population includes all participants who were randomized
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Remdesivir
Number analyzed (Participants) | 521 | 541
percentage of participants
  Death at or before study Visit | 1 [1 to 3] | 1 [0 to 2]
  Hospitalized, on invasive mech. vent. or ECMO | 36 [32 to 40] | 28 [25 to 32]
  Hospitalized, on non-invasive vent./high flow O2 | 17 [14 to 21] | 16 [13 to 19]
  Hospitalized, requiring supplemental oxygen | 32 [29 to 37] | 37 [33 to 41]
  Hospitalized, not on O2, requiring ongoing care | 12 [9 to 15] | 13 [10 to 16]
  Hospitalized, not requiring O2, no longer req care | 0.4 [0 to 1] | 0.2 [0 to 1]
  Not hospitalized, limit on activities/req home O2 | 0 [0 to 1] | 0 [0 to 1]
  Not hospitalized, no limitations on activities | 0 [0 to 1] | 0.4 [0 to 1]
  No clinical status score reported - Hospitalized | 0 [0 to 1] | 0 [0 to 1]
  No clinical status score reported - Discharged | 0.2 [0 to 1] | 2 [1 to 4]
  No clinical status score reported - Discontinued | 1 [0 to 2] | 2 [1 to 4]

19. Secondary Outcome: Percentage of Participants at Each Clinical Status Using Ordinal Scale at Day 5
Description: as for outcome 17
Time Frame: Day 5
Population: The intent-to-treat (ITT) population includes all participants who were randomized
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Remdesivir
Number analyzed (Participants) | 521 | 541
percentage of participants
  Death at or before study Visit | 2 [1 to 4] | 2 [1 to 4]
  Hospitalized, on invasive mech. vent. or ECMO | 37 [33 to 41] | 28 [24 to 32]
  Hospitalized, on non-invasive vent./high flow O2 | 14 [12 to 18] | 12 [9 to 15]
  Hospitalized, requiring supplemental oxygen | 26 [23 to 30] | 28 [24 to 31]
  Hospitalized, not on O2, requiring ongoing care | 11 [8 to 13] | 15 [12 to 18]
  Hospitalized, not requiring O2, no longer req care | 1 [0 to 2] | 1 [0 to 2]
  Not hospitalized, limit on activities/req home O2 | 0 [0 to 1] | 0.2 [0 to 1]
  Not hospitalized, no limitations on activities | 0.2 [0 to 1] | 0 [0 to 1]
  No clinical status score reported - Hospitalized | 0 [0 to 1] | 0 [0 to 1]
  No clinical status score reported - Discharged | 7 [5 to 9] | 12 [9 to 15]
  No clinical status score reported - Discontinued | 2 [1 to 3] | 3 [2 to 5]

20. Secondary Outcome: Percentage of Participants at Each Clinical Status Using Ordinal Scale at Day 8
Description: as for outcome 17
Time Frame: Day 8
Population: The intent-to-treat (ITT) population includes all participants who were randomized
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Remdesivir
Number analyzed (Participants) | 521 | 541
percentage of participants
  Death at or before study Visit | 7 [5 to 9] | 3 [2 to 5]
  Hospitalized, on invasive mech. vent. or ECMO | 33 [29 to 37] | 24 [21 to 28]
  Hospitalized, on non-invasive vent./high flow O2 | 9 [7 to 12] | 9 [7 to 12]
  Hospitalized, requiring supplemental oxygen | 15 [13 to 19] | 17 [14 to 21]
  Hospitalized, not on O2, requiring ongoing care | 10 [8 to 13] | 11 [9 to 14]
  Hospitalized, not requiring O2, no longer req care | 1 [1 to 3] | 1 [1 to 3]
  Not hospitalized, limit on activities/req home O2 | 0 [0 to 1] | 0.2 [0 to 1]
  Not hospitalized, no limitations on activities | 0.2 [0 to 1] | 0 [0 to 1]
  No clinical status score reported - Hospitalized | 0 [0 to 1] | 0.4 [0 to 1]
  No clinical status score reported - Discharged | 22 [19 to 26] | 30 [27 to 34]
  No clinical status score reported - Discontinued | 2 [1 to 3] | 4 [2 to 5]

21. Secondary Outcome: Percentage of Participants at Each Clinical Status Using Ordinal Scale at Day 11
Description: as for outcome 17
Time Frame: Day 11
Population: The intent-to-treat (ITT) population includes all participants who were randomized
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Remdesivir
Number analyzed (Participants) | 521 | 541
percentage of participants
  Death at or before study Visit | 8 [6 to 11] | 4 [3 to 6]
  Hospitalized, on invasive mech. vent. or ECMO | 28 [25 to 32] | 22 [19 to 26]
  Hospitalized, on non-invasive vent./high flow O2 | 7 [5 to 10] | 6 [4 to 8]
  Hospitalized, requiring supplemental oxygen | 13 [10 to 16] | 11 [9 to 14]
  Hospitalized, not on O2, requiring ongoing care | 6 [5 to 9] | 7 [5 to 9]
  Hospitalized, not requiring O2, no longer req care | 2 [1 to 4] | 2 [1 to 4]
  Not hospitalized, limit on activities/req home O2 | 0.4 [0 to 1] | 0.4 [0 to 1]
  Not hospitalized, no limitations on activities | 0.2 [0 to 1] | 0 [0 to 1]
  No clinical status score reported - Hospitalized | 0 [0 to 1] | 0 [0 to 1]
  No clinical status score reported - Discharged | 33 [29 to 37] | 44 [40 to 48]
  No clinical status score reported - Discontinued | 2 [1 to 4] | 4 [3 to 6]

22. Secondary Outcome: Percentage of Participants at Each Clinical Status Using Ordinal Scale at Day 15
Description: as for outcome 17
Time Frame: Day 15
Population: The intent-to-treat (ITT) population includes all participants who were randomized
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Remdesivir
Number analyzed (Participants) | 521 | 541
percentage of participants
  Death at or before study Visit | 11 [9 to 14] | 6 [5 to 9]
  Hospitalized, on invasive mech. vent. or ECMO | 22 [19 to 26] | 15 [13 to 19]
  Hospitalized, on non-invasive vent./high flow O2 | 4 [3 to 6] | 4 [3 to 6]
  Hospitalized, requiring supplemental oxygen | 11 [9 to 14] | 10 [8 to 13]
  Hospitalized, not on O2, requiring ongoing care | 6 [5 to 9] | 7 [5 to 9]
  Hospitalized, not requiring O2, no longer req care | 2 [1 to 3] | 3 [2 to 4]
  Not hospitalized, limit on activities/req home O2 | 17 [14 to 21] | 19 [16 to 22]
  Not hospitalized, no limitations on activities | 22 [19 to 26] | 29 [25 to 33]
  No clinical status score reported - Hospitalized | 0 [0 to 1] | 0 [0 to 1]
  No clinical status score reported - Discharged | 2 [1 to 3] | 2 [1 to 4]
  No clinical status score reported - Discontinued | 3 [2 to 4] | 5 [3 to 7]

23. Secondary Outcome: Percentage of Participants at Each Clinical Status Using Ordinal Scale at Day 22
Description: as for outcome 17
Time Frame: Day 22
Population: The intent-to-treat (ITT) population includes all participants who were randomized
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Remdesivir
Number analyzed (Participants) | 521 | 541
percentage of participants
  Death at or before study Visit | 13 [10 to 16] | 9 [7 to 12]
  Hospitalized, on invasive mech. vent. or ECMO | 14 [12 to 18] | 9 [7 to 12]
  Hospitalized, on non-invasive vent./high flow O2 | 2 [1 to 4] | 2 [1 to 4]
  Hospitalized, requiring supplemental oxygen | 8 [6 to 11] | 5 [4 to 8]
  Hospitalized, not on O2, requiring ongoing care | 5 [4 to 8] | 6 [4 to 8]
  Hospitalized, not requiring O2, no longer req care | 1 [0 to 2] | 1 [1 to 3]
  Not hospitalized, limit on activities/req home O2 | 18 [15 to 22] | 19 [16 to 23]
  Not hospitalized, no limitations on activities | 32 [29 to 37] | 39 [35 to 43]
  No clinical status score reported - Hospitalized | 0 [0 to 1] | 0 [0 to 1]
  No clinical status score reported - Discharged | 2 [1 to 4] | 3 [2 to 5]
  No clinical status score reported - Discontinued | 4 [2 to 6] | 6 [4 to 8]
  Completed study without reporting score | 0 [0 to 1] | 0.2 [0 to 1]

24. Secondary Outcome: Percentage of Participants at Each Clinical Status Using Ordinal Scale at Day 29
Description: as for outcome 17
Time Frame: Day 29
Population: The intent-to-treat (ITT) population includes all participants who were randomized
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Remdesivir
Number analyzed (Participants) | 521 | 541
percentage of participants
  Death at or before study Visit | 15 [12 to 18] | 11 [8 to 14]
  Hospitalized, on invasive mech. vent. or ECMO | 9 [7 to 11] | 6 [4 to 8]
  Hospitalized, on non-invasive vent./high flow O2 | 2 [1 to 3] | 1 [0 to 2]
  Hospitalized, requiring supplemental oxygen | 4 [3 to 6] | 4 [3 to 6]
  Hospitalized, not on O2, requiring ongoing care | 3 [2 to 5] | 3 [2 to 5]
  Hospitalized, not requiring O2, no longer req care | 1 [0 to 2] | 1 [0 to 2]
  Not hospitalized, limit on activities/req home O2 | 19 [16 to 23] | 20 [17 to 23]
  Not hospitalized, no limitations on activities | 36 [32 to 41] | 46 [42 to 50]
  No clinical status score reported - Hospitalized | 0.2 [0 to 1] | 0 [0 to 1]
  No clinical status score reported - Discharged | 3 [2 to 5] | 1 [1 to 3]
  No clinical status score reported - Discontinued | 5 [3 to 7] | 7 [5 to 9]
  Completed study without reporting score | 3 [2 to 4] | 2 [1 to 4]

25. Secondary Outcome: Percentage of Participants Reporting Grade 3 and 4 Clinical and/or Laboratory Adverse Events (AEs)
Description: Grade 3 AEs are defined as events that interrupt usual activities of daily living, or significantly affects clinical status, or may require intensive therapeutic intervention. Severe events are usually incapacitating. Grade 4 AEs are defined as events that are potentially life threatening.
Time Frame: Day 1 through Day 29
Population: The safety population includes all participants with available data post baseline, analyzed as treated.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Remdesivir
Number analyzed (Participants) | 516 | 532
percentage of participants | 57 [52.8 to 61.5] | 51 [47.0 to 55.6]
Statistical Analysis 1: Comparison: Placebo vs Remdesivir; Test type: Superiority; p = 0.058, Barnard's Exact Test

26. Secondary Outcome: Percentage of Participants Reporting Serious Adverse Events (SAEs)
Description: An SAE is defined as an AE or suspected adverse reaction is considered serious if, in the view of either the investigator or the sponsor, it results in death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect.
Time Frame: Day 1 through Day 29
Population: The safety population includes all participants with available data post baseline, analyzed as treated.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Remdesivir
Number analyzed (Participants) | 516 | 532
percentage of participants | 32 [27.7 to 35.7] | 24 [20.9 to 28.3]
Statistical Analysis 1: Comparison: Placebo vs Remdesivir; Test type: Superiority; p = 0.010, Barnard's Exact Test

27. Secondary Outcome: Percentage of Participants Discontinued or Temporarily Suspended From Investigational Therapeutics
Description: Participants may have been discontinued from investigational therapeutics due to discharge or death. The halting or slowing of the infusion for any reason was collected, as was missed doses in the series of 10 doses.
Time Frame: Day 1 through Day 10
Population: The intent-to-treat (ITT) population includes all participants who were randomized
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Remdesivir
Number analyzed (Participants) | 521 | 541
percentage of participants
  Discontinued due to discharge | 30 [26 to 34] | 41 [37 to 45]
  Discontinued due to death | 4 [2 to 6] | 3 [2 to 5]
  Any infusions halted or slowed | 2 [1 to 4] | 2 [1 to 4]
  Missed any maintenance dose | 21 [18 to 25] | 16 [13 to 19]

28. Secondary Outcome: Duration of Hospitalization
Description: Duration of hospitalization was determined two ways. The first includes imputations for participants who died. The second method is restricted to participants who did not die.
Time Frame: Day 1 through Day 29
Population: The intent-to-treat (ITT) population includes all participants who were randomized
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Placebo | Remdesivir
Number analyzed (Participants) | 521 | 541
Days
  Including imputation for participants who died | 17 [8 to 28] | 12 [6 to 28]
  Restricted to participants who did not die: number analyzed (Participants) | 443 | 480
  Restricted to participants who did not die | 14 [7 to 27] | 10 [5 to 21]

29. Secondary Outcome: Duration of New Non-invasive Ventilation or High Flow Oxygen Use
Description: Duration of new non-invasive ventilation or high flow oxygen use was measured in days among participants who were not on non-invasive ventilation or high-flow oxygen use at baseline, determined two ways. The first includes imputations for participants who died. The second method is restricted to participants who did not die
Time Frame: Day 1 through Day 29
Population: The analysis population is restricted to randomized participants who were not on non-invasive ventilation or high-flow oxygen at baseline but who subsequently required non-invasive or high-flow oxygen.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Placebo | Remdesivir
Number analyzed (Participants) | 64 | 52
Days
  Including imputations for participants who died | 4 [2 to 23.5] | 3 [1 to 10.5]
  Among participants who did not die: number analyzed (Participants) | 50 | 43
  Among participants who did not die | 3 [2 to 6] | 3 [1 to 6]

30. Secondary Outcome: Duration of New Oxygen Use
Description: Duration of new oxygen use was measured in days among participants who were not on oxygen at baseline, determined two ways. The first includes imputations for participants who died. The second method is restricted to participants who did not die
  .
Time Frame: Day 1 through Day 29
Population: The analysis population is restricted to randomized participants who were not on oxygen at baseline but who subsequently required oxygen.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Placebo | Remdesivir
Number analyzed (Participants) | 28 | 27
Days
  Including imputations for participants who died | 5.5 [1 to 15] | 4 [2 to 12]
  Among participants who did not die: number analyzed (Participants) | 25 | 24
  Among participants who did not die | 3 [1 to 13] | 3.5 [2 to 5.5]

31. Secondary Outcome: Duration of New Ventilator or Extracorporeal Membrane Oxygenation (ECMO) Use
Description: Duration of new ventilator or ECMO use was measured in days among participants who were not on a ventilator or ECMO at baseline, determined two ways. The first includes imputations for participants who died. The second method is restricted to participants who did not die
Time Frame: Day 1 through Day 29
Population: The analysis population is restricted to randomized participants not on a ventilator or ECMO at baseline but who subsequently required a ventilator or ECMO.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Placebo | Remdesivir
Number analyzed (Participants) | 82 | 52
Days
  Including imputations for participants who died | 23 [12 to 28] | 21.5 [9 to 28]
  Among participants who did not die: number analyzed (Participants) | 57 | 39
  Among participants who did not die | 16 [9 to 24] | 14 [5 to 26]

32. Secondary Outcome: Percentage of Participants Requiring New Non-invasive Ventilation or High-flow Oxygen Use
Description: New non-invasive ventilation or high-flow oxygen use was determined as the percentage of subject not on non-invasive ventilation or high-flow oxygen at baseline.
Time Frame: Day 1 through Day 29
Population: The analysis population is restricted to randomized participants who were not on non-invasive or high-flow oxygen at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Remdesivir
Number analyzed (Participants) | 266 | 307
percentage of participants | 24 [19 to 30] | 17 [13 to 22]

33. Secondary Outcome: Percentage of Participants Requiring New Oxygen Use
Description: The percentage of participants requiring new oxygen use was determined as the percentage of participants not requiring oxygen at baseline
Time Frame: Day 1 through Day 29
Population: The analysis population is restricted to randomized participants not requiring oxygen at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Remdesivir
Number analyzed (Participants) | 63 | 75
percentage of participants | 44 [33 to 57] | 36 [26 to 47]

34. Secondary Outcome: Percentage of Participants Requiring New Ventilator or Extracorporeal Membrane Oxygenation (ECMO) Use
Description: The percentage of participants requiring new ventilator or ECMO use was determined as the percentage not on a ventilator or ECMO at baseline
Time Frame: Day 1 through Day 29
Population: The analysis population is restricted to randomized participants not on a ventilator or ECMO at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Remdesivir
Number analyzed (Participants) | 364 | 402
percentage of participants | 23 [19 to 27] | 13 [10 to 17]

35. Secondary Outcome: Mean Change in the Ordinal Scale
Description: The ordinal scale is an assessment of the clinical status at the first assessment of a given study day. The scale is as follows: 8) Death; 7) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 6) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 5) Hospitalized, requiring supplemental oxygen; 4) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 3) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 2) Not hospitalized, limitation on activities and/or requiring home oxygen; 1) Not hospitalized, no limitations on activities. A positive change indicates a worsening and a negative change is an improvement.
Time Frame: Day 1, 3, 5, 8, 11, 15, 22, and 29
Population: The intent-to-treat (ITT) population includes all participants who were randomized reporting a clinical score. Missing values were imputed using Last Observation Carried Forward. Clinical scores of 8 were carried forward from the date of death for participants who died.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Remdesivir
Number analyzed (Participants) | 518 | 533
units on a scale
  Day 3 | 0.2 (0.6) | 0.1 (0.6)
  Day 5 | 0.1 (0.9) | 0.0 (0.8)
  Day 8 | 0.0 (0.1) | -0.2 (1.0)
  Day 11 | -0.1 (1.3) | -0.3 (1.1)
  Day 15 | -1.4 (2.3) | -1.9 (2.1)
  Day 22 | -1.9 (2.5) | -2.4 (2.2)
  Day 29 | -2.3 (2.6) | -2.7 (2.3)

36. Secondary Outcome: 14-day Participant Mortality
Description: The mortality rate was determined as the proportion of participants who died by study Day 15.
Time Frame: Day 1 through Day 15
Population: The ITT population consists of all participants as randomized.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Placebo | Remdesivir
Number analyzed (Participants) | 521 | 541
Proportion of participants | 0.12 [0.09 to 0.15] | 0.07 [0.05 to 0.09]

37. Secondary Outcome: 29-day Participant Mortality
Description: The mortality rate was determined as the proportion of participants who died by study Day 29.
Time Frame: Day 1 through Day 29
Population: The ITT population includes all participants as randomized
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Placebo | Remdesivir
Number analyzed (Participants) | 521 | 541
Proportion of participants | 0.15 [0.12 to 0.19] | 0.11 [0.09 to 0.15]

38. Secondary Outcome: Time to an Improvement by at Least One Category Using an Ordinal Scale
Description: The ordinal scale is an assessment of the clinical status at the first assessment of a given study day. The scale is as follows: 8) Death; 7) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 6) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 5) Hospitalized, requiring supplemental oxygen; 4) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 3) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 2) Not hospitalized, limitation on activities and/or requiring home oxygen; 1) Not hospitalized, no limitations on activities. Time to improvement by at least one category was determined for each participant
Time Frame: Day 1 through Day 29
Population: The ITT population includes all participants as randomized
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo | Remdesivir
Number analyzed (Participants) | 521 | 541
Days | 9 [8 to 11] | 7 [6 to 8]
Statistical Analysis 1: Comparison: Placebo vs Remdesivir; Test type: Superiority; p = 0.002, Log Rank; Cox Proportional Hazard = 1.23, 95% CI 2-sided [1.08 to 1.41]

39. Secondary Outcome: Time to an Improvement of at Least Two Categories Using an Ordinal Scale
Description: The ordinal scale is an assessment of the clinical status at the first assessment of a given study day. The scale is as follows: 1) Death; 2) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 3) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4) Hospitalized, requiring supplemental oxygen; 5) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 6) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 7) Not hospitalized, limitation on activities and/or requiring home oxygen; 8) Not hospitalized, no limitations on activities. Time to improvement by at least two categories was determined for each participant
Time Frame: Day 1 through Day 29
Population: The ITT population includes all participants as randomized
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo | Remdesivir
Number analyzed (Participants) | 521 | 541
Days | 14 [13 to 15] | 11 [10 to 13]
Statistical Analysis 1: Comparison: Placebo vs Remdesivir; Test type: Superiority; p < 0.001, Log Rank; Cox Proportional Hazard = 1.29, 95% CI 2-sided [1.12 to 1.48]

40. Secondary Outcome: Time to Discharge or to a NEWS of 2 or Less and Maintained for 24 Hours, Whichever Occurs First
Description: The NEW score has demonstrated an ability to discriminate patients at risk of poor outcomes. This score is based on 7 clinical parameters (respiration rate, oxygen saturation, any supplemental oxygen, temperature, systolic blood pressure, heart rate, level of consciousness). The NEW Score is being used as an efficacy measure. The minimum score is 0, representing the better outcome, and the maximum value is 19, representing the worse outcome. The time to discharge or a NEWS of less than or equal to 2 was determined for each participant.
Time Frame: Day 1 through Day 29
Population: The ITT population includes all participants as randomized.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo | Remdesivir
Number analyzed (Participants) | 521 | 541
Days | 12 [10 to 15] | 8 [7 to 9]
Statistical Analysis 1: Comparison: Placebo vs Remdesivir; Test type: Superiority; p < 0.001, Log Rank; Cox Proportional Hazard = 1.27, 95% CI 2-sided [1.10 to 1.46]

41. Primary Outcome: Time to Recovery by Race
Description: as for outcome 1
Time Frame: Day 1 through Day 29
Population: The intent-to-treat (ITT) population includes all participants who were randomized
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo | Remdesivir
Number analyzed (Participants) | 521 | 541
Days
  Asian: number analyzed (Participants) | 56 | 79
  Asian | 12.0 [9.0 to 15.0] | 11.0 [9.0 to 15.0]
  Black or African American: number analyzed (Participants) | 117 | 109
  Black or African American | 15.0 [10.0 to 21.0] | 10.0 [7.0 to 16.0]
  White: number analyzed (Participants) | 287 | 279
  White | 15.0 [12.0 to 19.0] | 9.0 [8.0 to 12.0]
  Other: number analyzed (Participants) | 61 | 74
  Other | 24.0 [15.0 to NA] — A large number of participants at the median estimate resulted in little variability at the 50th percentile and the methodology described by Klein and Moeschberger (1997) was unable to compute an upper confidence limit. | 9.0 [6.0 to 14.0]
Statistical Analysis 1: Comparison: Placebo vs Remdesivir; This analysis is for Asian participants; Test type: Superiority; Cox Proportional Hazard = 1.07, 95% CI 2-sided [0.73 to 1.58]
Statistical Analysis 2: Comparison: Placebo vs Remdesivir; This analysis is for Black or African American participants; Test type: Superiority; Cox Proportional Hazard = 1.25, 95% CI 2-sided [0.91 to 1.72]
Statistical Analysis 3: Comparison: Placebo vs Remdesivir; This analysis is for White participants; Test type: Superiority; Cox Proportional Hazard = 1.29, 95% CI 2-sided [1.06 to 1.57]
Statistical Analysis 4: Comparison: Placebo vs Remdesivir; This analysis is for Race of Other participants; Test type: Superiority; Cox Proportional Hazard = 1.68, 95% CI 2-sided [1.10 to 2.58]

42. Primary Outcome: Time to Recovery by Ethnicity
Description: as for outcome 1
Time Frame: Day 1 through Day 29
Population: The intent-to-treat (ITT) population includes all participants who were randomized and for whom Ethnicity was reported
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo | Remdesivir
Number analyzed (Participants) | 489 | 516
Days
  Not Hispanic or Latino: number analyzed (Participants) | 373 | 382
  Not Hispanic or Latino | 15.0 [13.0 to 18.0] | 10.0 [8.0 to 12.0]
  Hispanic or Latino: number analyzed (Participants) | 116 | 134
  Hispanic or Latino | 12.5 [9.0 to 22.0] | 10.0 [7.0 to 14.0]
Statistical Analysis 1: Comparison: Placebo vs Remdesivir; This analysis is for Not Hispanic or Latino participants; Test type: Superiority; Cox Proportional Hazard = 1.31, 95% CI 2-sided [1.10 to 1.55]
Statistical Analysis 2: Comparison: Placebo vs Remdesivir; This analysis is for Hispanic or Latino participants; Test type: Superiority; Cox Proportional Hazard = 1.28, 95% CI 2-sided [0.94 to 1.73]

43. Primary Outcome: Time to Recovery by Sex
Description: as for outcome 1
Time Frame: Day 1 through Day 29
Population: The intent-to-treat (ITT) population includes all participants who were randomized
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo | Remdesivir
Number analyzed (Participants) | 521 | 541
Days
  Male: number analyzed (Participants) | 332 | 352
  Male | 15.0 [12.0 to 19.0] | 9.0 [8.0 to 12.0]
  Female: number analyzed (Participants) | 189 | 189
  Female | 15.0 [12.0 to 19.0] | 10.0 [8.0 to 13.0]
Statistical Analysis 1: Comparison: Placebo vs Remdesivir; This analysis is for Male participants; Test type: Superiority; Cox Proportional Hazard = 1.30, 95% CI 2-sided [1.09 to 1.56]
Statistical Analysis 2: Comparison: Placebo vs Remdesivir; This analysis is for Female participants; Test type: Superiority; Cox Proportional Hazard = 1.31, 95% CI 2-sided [1.03 to 1.66]

ADVERSE EVENTS:
Time Frame: Grade 3 and 4 serious and non-serious adverse events were collected for 29 days after the first dose. Laboratory values were systematically assessed at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29.
Description: Given the nature of severity of the underlying illness, participants were expected to have many symptoms and abnormalities in vital signs and laboratory values. All Grade 3 and 4 AEs were captured as AEs in this trial. In addition, any Grade 2 or higher, suspected drug-related hypersensitivity reaction was to be reported as an AE in this trial. All cause mortality was calculated for the ITT population, while SAEs and AEs reflect the as treated population.
Arm/Group | Placebo | Remdesivir
All-Cause Mortality (participants affected / at risk) | 77/521 | 59/541
Serious Adverse Events (participants affected / at risk) | 163/516 | 131/532
Other Adverse Events (participants affected / at risk) | 295/516 | 276/532
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=516) | Remdesivir (N=532)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 7 (7) | 10 (10)
Atrial fibrillation (Cardiac disorders) | 1 (2) | 5 (6)
Cardio-respiratory arrest (Cardiac disorders) | 3 (3) | 1 (1)
Myocardial infarction (Cardiac disorders) | 4 (4) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 3 (3) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 2 (2) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 3 (3) | 5 (5)
Pyrexia (General disorders) | 2 (2) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Ischaemic hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 15 (15) | 8 (8)
COVID-19 (Infections and infestations) | 5 (5) | 2 (2)
Bacteraemia (Infections and infestations) | 2 (2) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Catheter bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 0 (0) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 2 (3) | 5 (5)
Haemoglobin decreased (Investigations) | 2 (2) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 3 (3)
Seizure (Nervous system disorders) | 1 (1) | 2 (2)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic transformation stroke (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Intensive care unit acquired weakness (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 12 (12) | 7 (7)
Renal failure (Renal and urinary disorders) | 5 (5) | 2 (2)
Renal impairment (Renal and urinary disorders) | 3 (3) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 58 (59) | 35 (36)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 8 (8)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 6 (6)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 7 (7)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Endotracheal intubation (Surgical and medical procedures) | 9 (9) | 6 (6)
Mechanical ventilation (Surgical and medical procedures) | 3 (3) | 1 (1)
Hypotension (Vascular disorders) | 7 (7) | 4 (4)
Shock (Vascular disorders) | 4 (4) | 5 (5)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Embolism venous (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=516) | Remdesivir (N=532)
Glomerular filtration rate decreased (Investigations) | 74 (81) | 55 (59)
Haemoglobin decreased (Investigations) | 62 (69) | 48 (51)
Lymphocyte count decreased (Investigations) | 54 (63) | 44 (56)
Anaemia (Blood and lymphatic system disorders) | 52 (58) | 42 (52)
Pyrexia (General disorders) | 32 (37) | 38 (52)
Hyperglycaemia (Metabolism and nutrition disorders) | 34 (43) | 34 (36)
Blood creatinine increased (Investigations) | 36 (41) | 31 (33)
Blood glucose increased (Investigations) | 27 (31) | 39 (45)
Aspartate aminotransferase increased (Investigations) | 33 (35) | 18 (19)
Lymphopenia (Blood and lymphatic system disorders) | 30 (34) | 13 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2020-04-02): https://cdn.clinicaltrials.gov/large-docs/05/NCT04280705/Prot_001.pdf
  • Statistical Analysis Plan (2020-05-29): https://cdn.clinicaltrials.gov/large-docs/05/NCT04280705/SAP_002.pdf
  • Informed Consent Form (2020-03-04): https://cdn.clinicaltrials.gov/large-docs/05/NCT04280705/ICF_000.pdf